CLINICAL TRIAL: NCT04810858
Title: Modeling the Effects of Chronic Marijuana Use on Neuroinflammation and HIV-related Neuronal Injury
Acronym: CHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00098474; R01DA052827 (NIH)
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-04

CONDITIONS: Cannabis; HIV; Inflammation; Cognition; Neuroimaging
MeSH Terms: conditions — Marijuana Abuse; Inflammation | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of 4 study groups: HIV+ marijuana user, HIV+ non-drug user, HIV- marijuana users, and HIV- non-drug user
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIV+ marijuana user (Other): Participants with HIV who report marijuana use
  Interventions: Other: Multimodal, multi-parametric MRI; Other: Immune and cytokine profiling; Behavioral: Neuropsychological testing
- HIV+ non-drug user (Other): Participants with HIV who report no drug use
  Interventions: Other: Multimodal, multi-parametric MRI; Other: Immune and cytokine profiling; Behavioral: Neuropsychological testing
- HIV- marijuana user (Other): Participants without HIV who report marijuana use
  Interventions: Other: Multimodal, multi-parametric MRI; Other: Immune and cytokine profiling; Behavioral: Neuropsychological testing
- HIV- non-drug user (Other): Participants without HIV who report no drug use
  Interventions: Other: Multimodal, multi-parametric MRI; Other: Immune and cytokine profiling; Behavioral: Neuropsychological testing

INTERVENTIONS:
Other: Multimodal, multi-parametric MRI — The investigators will use multimodal, multi-parametric sequences to investigate neuroinflammatory and neurodegenerative processes in vivo. Participants will be assessed three times over 2 years.
Other: Immune and cytokine profiling — Blood samples will be collected for immune and cytokine profiling. Participants will be assessed three times over 2 years.
Behavioral: Neuropsychological testing — Participants will have neuropsychological testing three times over 2 years.

SUMMARY:
This study applies a hypothesis-driven approach to examine the effects of chronic marijuana use on HIV-associated inflammation and its subsequent impacts on central nervous system function, with the goal of identifying the mechanisms through which cannabinoids modulate neurological disorders and other comorbidities in persons with HIV.

ELIGIBILITY:
Inclusion Criteria:

* verified HIV status
* Current marijuana use (MJ+ groups only)
* No current marijuana use (MJ- groups only)
* current engagement in HIV care (HIV+ participants only)
* receipt of cART as first-line of treatment (HIV+ participants only)
* stable cART regimen (HIV+ participants only)
* undetectable HIV RNA viral load for >1 year (HIV+ participants only)

Exclusion Criteria:

* Lifetime abuse for any illicit drug other than marijuana
* <9th grade education; illiteracy or lack of fluency in English
* history of moderate or severe head trauma
* unstable or serious neurological disorders
* severe mental illness
* systemic autoimmune diseases
* immunotherapy
* MRI contraindications

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in neurocognitive function as measured by neuropsychological battery | baseline, 1-year follow-up, and 2-year follow-up
  The neuropsychological testing battery assesses 7 cognitive domains with 3-4 tests per domain. Raw scores from each test will be converted to demographically adjusted standard scores, called T-scores using up-to-date US normative data. A T-score of 50 is considered the normative mean, and each 10-point deviation is equivalent to 1 standard deviation. The minimum possible T-score is 0 and the maximum is 100, with higher scores meaning better neurocognitive function. The average T-score for all tests in a domain will be the domain T-score, and the average of all domain T-scores will be the global T-score. T-scores will serve as the primary continuous measure because they capture the full range of cognitive function.
Change in neuronal integrity as measured by N-acetyl aspartate (NAA) | baseline, 1-year follow-up, and 2-year follow-up
  NAA will be measured using Echo-planar spectroscopic imaging. Lower NAA is associated with less neuronal integrity. NAA units of measure is parts per million.
Change in neuronal-glial interaction as measured by Glutamate + glutamine (GLX) | baseline, 1-year follow-up, and 2-year follow-up
  GLX will be measured using Echo-planar spectroscopic imaging. Lower GLX is indicative of less neuronal-glial interactions. GLX units of measure is parts per million.
Change in axonal loss and injury as measured by axonal diffusivity (AD) | baseline, 1-year follow-up, and 2-year follow-up
  AD will be measured using diffusion-weighted imaging. Lower axonal diffusivity is associated with more axonal loss and injury. The unit of measure for AD is micrometer^2/millisecond.
Change in demyelination or dysmyelination as measured by radial diffusivity (RD) | baseline, 1-year follow-up, and 2-year follow-up
  RD will be measured using diffusion-weighted imaging. Higher radial diffusivity is associated with more demyelination and dysmyelination. The unit of measure for RD is micrometer^2/millisecond.
Change in overall white matter integrity as measured by fractional anisotropy (FA) | baseline, 1-year follow-up, and 2-year follow-up
  FA will be measured using diffusion-weighted imaging. Higher FA is associated with higher overall white matter integrity. FA is a scalar value between 0 and 1.
Change in inflammation-related cellularity as measured by restricted fraction (RF) | baseline, 1-year follow-up, and 2-year follow-up
  RF will be measured using diffusion-weighted imaging. Higher restricted fraction is associated with higher inflammation-related cellularity. The unit of measure for RF is micrometer^2/millisecond.
Change in extracellular tissue edema as measured by non-restricted fraction (NF) | baseline, 1-year follow-up, and 2-year follow-up
  NF will be measured using diffusion-weighted imaging. Lower non-restricted fraction is associated with increased extracellular tissue edema. The unit of measure for NF is micrometer^2/millisecond.
Change in gray matter as measured by cortical area and thickness and cortical and subcortical volume | baseline, 1-year follow-up, and 2-year follow-up
  Cortical areas and thickness and cortical and subcortical volume will be measured using T1-weighted imaging. Lower gray matter is associated with decreased cognitive function and is a marker of neurodegenerative disease. Cortical area, thickness, and volume units of measure are in millimeter^2. Subcortical volume units of measure are in millimeter^3.
Change in white matter integrity as measured by white matter tract streamline count | baseline, 1-year follow-up, and 2-year follow-up
  White matter tract streamline count will be measured using diffusion-weighted imaging. Lower white matter tract streamline count is associated with lower white matter integrity. The unit of measure for white matter tract streamline count is the total number of streamlines within a white matter tract.
Change in axonal damage was measured by neurofilament light (NfL) protein | baseline, 1-year follow-up, and 2-year follow-up
  NfL will be measured using blood serum and processed using an ultrasensitive immunoassay. Higher NfL is associated with more axonal damage. NfL protein units of measure are in picogram/milliliter^-1.

CONTACTS AND LOCATIONS:
Overall Officials: Christina S Meade, PhD, Principal Investigator — Duke University
Locations (1):
- Biotech Place, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Any guidelines, protocols, and operating procedures generated will be made freely available. The investigators will make the data and associated documentation available to users under a data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The investigators will lock the data until the primary analyses are completed and accepted for publication, after which the investigators will make the data as widely available as possible.
Access Criteria: Data sharing agreements will include: (1) a commitment to acknowledge the sources of the data and conform to the terms and conditions under which they accessed it, (2) a commitment to use the data only for research purposes and not to identify any individual participant, (3) a commitment to securing the data using appropriate computer technology, and (4) a commitment to destroying or returning the data after analyses are completed.